CLINICAL TRIAL: NCT01730066
Title: Probiotics for Reduction of Pathogenic Bacteria in Connection With Advanced Surgery in the Mouth, the Oropharynx, and on the Neck
Brief Title: Probiotics Against Pathogenic Bacteria in Advanced ENT-Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ProOncENT
Record Dates: First submitted 2012-11-08; First posted 2012-11-21 (Estimated); Last update posted 2020-10-12 (Actual); Status verified 2020-10

CONDITIONS: Advanced ENT Surgery; Microbiological Flora in the Oropharynx and Lower Airways
Keywords: Probiotics; Pathogenic enteric bacteria; Oropharyngeal flora; CRP; WBC
MeSH Terms: interventions — maltodextrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotics (Experimental): Patients will gurgle and swallow a mixture of probiotic bacteria preoperatively and given the same study product enterally postoperatively
  Interventions: Dietary Supplement: L. plantarum 299 and L. plantarum 299v (+maltodextrin)
- Control (No Intervention): No intervention.What has been the standard procedure so far

INTERVENTIONS:
Dietary Supplement: L. plantarum 299 and L. plantarum 299v (+maltodextrin) — Patients will be given a mixture of maltodextrin ( a starch product often used i alimentary products) and two strains of probiotic bacteria ( L. plantarum 299 and L. plantarum 299v ) dissolved in water. They will gurgle and swallow the suspension from the day before surgery. Postoperatively they will be given the probiotic mixture via a nasogastric tubing twice a day and when the responsible surgeon find it suitable also orally as described above. When they can swallow no study product is given through the nasogastric tube.
  Patients randomized 1:1 between groups
  Arms: Probiotics

SUMMARY:
Surgery in the mouth and oropharynx is performed in an area colonised by bacteria non-pathogenic and pathogenic.

Antibiotics are used regularly resulting in disturbances in the intestinal microbiological flora and consequently diarrhoea that can be troublesome. The use of antibiotics throughout the hospital stay for these difficult cases represent a risk of development of resistant strains.

Most of the patients have cancer diagnoses and have radiation therapy before surgery. This increases the risk of the patients having pathogenic bacteria normally present in the lower GI-tract.

The investigators have shown for ICU patients that treatment with probiotics reduces the number of emerging enteral bacteria in the oropharynx and now the investigators will perform an adjusted procedure for patients planned for large ear, nose, and throat (ENT) surgery.

Patients will preoperatively gurgle a suspension of probiotics and then swallow the preparation.

Postoperatively the probiotics is given enterally and a eventually by mouth again.

Cultures will be taken from the oropharynx and tracheal secretions and the results will be compared

DETAILED DESCRIPTION:
Longer surgical procedures require intubation and there is a potential risk of contaminating the lower airways with pathogenic bacteria from the mouth and oropharynx.

Surgery including the mouth and the oropharynx is performed in an area that is colonised by hundreds of different bacterial species. In the healthy person there is a balance between the different microbes and possible pathogens are kept under control.

Patients that are subject to surgery in the mouth, oropharynx or neck area, most often have cancer diagnoses. Preoperative treatment (mostly radiation) is done in most cases resulting in a changed spectrum of bacteria in the mouth and oropharynx. Due to lowered appetite increased difficulties to eat, in combination with cancer diagnosis, there is also a change in cranial direction of the microbiological gut flora resulting in the presence of pathogens such as Gram-negative bacteria. Those species may result in troublesome infections in the postoperative period.

With healthy people pathogenic bacteria originating from the gastro/intestinal canal are seldom found in the oropharynx, but those do occur among many patients.

Antibiotics are used prophylactic and for more extensive surgery, as micro vascular procedures with free transplants of tissues, antibiotics are kept throughout the length of stay (LOS) in hospital. This results in an increased risk for the development of resistant bacteria and does result in changes in the GI flora in those patients. Diarrhoea occurs frequently and are troublesome for the patients For ICU patients we have seen a reduction of emerging enteric bacteria in patients given oral care with probiotics and this study will explore the possibility of the same kind of positive effects in patients due for extensive surgery performed during several hours.

Many of the patients will have a tracheostomy performed as part of the surgical procedure.

Patients will be randomised (1:1) to either no prophylaxis (standard procedure today) or to preparation with a probiotic suspension fro the day before surgery until discharge from hospital.

Preoperatively the patients will gurgle a suspension of probiotics and then swallow the preparation.

Postoperatively the probiotics is given enterally and a eventually when the responsible surgeon find it suitable by mouth again.

Cultures at inclusion, after intubation, and then on predefined days postoperatively to compare bacterial flora in the oropharynx and in tracheal secretions.

Infectious parameters will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Elective advanced and extensive ENT surgery
* Adult patients (≥ 18 years)
* Surgery requires general anesthesia and endotracheal intubation
* Length of anesthesia ≥ 1,5 hours
* Signed informed consent

Exclusion Criteria:

* Ongoing treatment requiring infection in the lower respiratory tract
* Chronic lung disease requiring oxygen treatment
* Known immune deficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Differences in pathogenic bacteria in the oropharynx | During hospitalization, anticipated mean time 12 days
  Emerging and resident bacteria will be compared for the cultures taken in the oropharynx and from tracheal secretions in connection to a surgical intervention and postoperatively

SECONDARY OUTCOMES:
White Blood Cell count | During hospital stay, expected mean LOS 12 days
  WBC taken pre-op and then on predefined days postoperatively
C Reactive Protein | Throughout the hospital stay, expected mean LOS 12 days
  CRP taken pre-op and then on predefined days postoperatively
Length of Hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 2-3 weeks
  Length of stay is recorded for the Hospital stay, and for those cases that have an extended post-operative period in the ICU, the length of the ICU stay will be recorded
Survival | Six months
  For participating patients the status of survival or non survival at days 28 and 180 (six months) will be recorded
Diarrhoea and obstipation | Throughout the hospital stay, expected mean LOS 12 days
  As ICU patients tend to display diarrhoea as well as obstipation the frequency and consistency of stools will be recorded.
  Probiotics are anticipated to stabilise bowel function

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Klarin, MD, PhD, Principal Investigator — Lund University Hospital
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Results will be published in a scientific journal

REFERENCES:
- [Background] Stjernquist-Desatnik A, Warfving H, Johansson ML. Persistence of Lactobacillus plantarum DSM 9843 on human tonsillar surface after oral administration in fermented oatmeal gruel. A pilot study. Acta Otolaryngol Suppl. 2000;543:215-9. doi: 10.1080/000164800454422. PMID 10909023
- [Background] Klarin B, Molin G, Jeppsson B, Larsson A. Use of the probiotic Lactobacillus plantarum 299 to reduce pathogenic bacteria in the oropharynx of intubated patients: a randomised controlled open pilot study. Crit Care. 2008;12(6):R136. doi: 10.1186/cc7109. Epub 2008 Nov 6. PMID 18990201
- See also: Provider of study product — http://www.probi.se